CLINICAL TRIAL: NCT07160998
Title: An Active Health-Based Comprehensive Study on Diabetes Management
Acronym: X Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li Huating (Other)
Responsible Party: Sponsor-Investigator, Li Huating, Shanghai 6th People's Hospital, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-122
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- X Life AI Lifestyle Guidance (Experimental): Personalized real-time lifestyle recommendations delivered via smartphone, tablet, etc., integrating glucose level and wearable data.
  Interventions: Other: Digital Lifestyle Therapeutic
- Standard Care (Active Comparator): Participants receive standard diabetes management including medications and lifestyle recommendations based on guidelines.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Other: Digital Lifestyle Therapeutic — Personalized real-time lifestyle recommendations are delivered via via smartphone, tablet, etc., integrating glucose level and wearable data.
  Arms: X Life AI Lifestyle Guidance
Behavioral: Standard Care — Participants receive standard diabetes management including medications and lifestyle recommendations based on guidelines.
  Arms: Standard Care

SUMMARY:
This randomized, open-label, multicenter trial evaluates the efficacy and safety of the AI-based lifestyle guidance system (X-Life) compared to standard care in adults with type 2 diabetes. X-Life integrates glucose level, wearable devices, and AI-driven decision models to provide personalized lifestyle recommendations. The primary endpoint is the percentage of time in glucose target range (TIR).

DETAILED DESCRIPTION:
Type 2 diabetes imposes a global health burden. Traditional care has limitations in accessibility, personalization, and long-term adherence. AI-driven digital therapeutics may overcome these barriers. X-Life is an innovative AI system providing individualized lifestyle guidance using glucose level and wearable data. User studies demonstrated usability and acceptability. This multicenter randomized controlled trial will rigorously test whether X-Life improves glycemic control compared with standard care, while also evaluating metabolic outcomes, patient-reported measures, and safety. The investigators designed this trial with the assistance of a digital twin-based clinical research system (termed X Town).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosed type 2 diabetes
* Stable medication regimen ≥ 3 months
* HbA1c 7-10%
* Smartphone access and ability to operate app
* Willing to wear CGM and activity tracker
* Able to provide informed consent

Exclusion Criteria:

* Insulin therapy
* Severe chronic/acute diabetic complications
* Early-onset diabetes (<40 years at diagnosis)
* Severe cardiovascular disease, uncontrolled hypertension, active liver disease, malignancy
* Severe psychiatric or cognitive disorders
* Allergy to CGM materials
* Planned surgery or long-term travel during study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2025-09-07 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Time in Range (TIR, %) | Run-in period (Day -7 to Day 0) and intervention period (Day 1 to Day 28)
  Percentage of glucose readings within 3.9-10 mmol/L measured by CGM

SECONDARY OUTCOMES:
Other CGM metrics | Run-in period (Day -7 to Day 0) and intervention period (Day 1 to Day 28)
  mean glucose, SD, CV, TAR (>10 mmol/L), TBR (<3.9 and <3.0 mmol/L), daytime/nighttime TIR, MAGE, MODD, AUC, etc.
Patient-reported outcomes | Baseline and 28 days
  Using DDS, DSCS, Self-Efficacy, WHO-5 scales, etc.
User Experience Score | At 28 days
  Evaluation in X Life group only. User experience will be assessed using a validated questionnaire covering usability, usefulness, satisfaction, and acceptability. Each item is rated on a 5-point Likert scale. Higher scores indicate better user experience.
Safety outcomes | Day 1-28 (intervention period)
  Number of participants with CGM-recorded or symptomatic hypoglycemia (<3.9 mmol/L). Number of participants experiencing any AE/SAE.
OGTT Glucose Concentration | Baseline and 28 days
  Plasma glucose at 0, 60, and 120 minutes during OGTT.
OGTT Insulin Concentration | Baseline and 28 days
  Serum insulin at 0, 60, and 120 minutes during OGTT.
OGTT C-peptide Concentration | Baseline and 28 days
  Serum C-peptide at 0, 60, and 120 minutes during OGTT.
Body Weight | Baseline and 28 days
  Body weight (kg) measured using digital scale.
Body Mass Index (BMI) | Baseline and 28 days
  Calculated as weight (kg) / height (m²).
Waist Circumference | Baseline and 28 days
  Measured at the midpoint between the lowest rib and iliac crest.
Hip Circumference | Baseline and 28 days
  Hip circumference measured at the widest part of the buttocks using a non-stretchable tape.
Thigh Circumference | Baseline and 28 days
  Mid-thigh circumference measured at the midpoint between the inguinal crease and the proximal border of the patella.
Systolic Blood Pressure | Baseline and 28 days
  Average of two seated measurements.
Diastolic Blood Pressure | Baseline and 28 days
  Average of two seated measurements.
Resting Heart Rate | Baseline and 28 days
  Measured by automated device after 5 minutes rest.
Blood Lipids | Baseline and 28 days
  Total cholesterol, LDL-C, HDL-C, and triglycerides.
Liver Function | Baseline and 28 days
  ALT, AST, GGT, etc.
Kidney Function | Baseline and 28 days
  Serum creatinine, eGFR, etc.
Inflammatory Markers | Baseline and 28 days
  C-reactive protein
Composite Psychological and Behavioral Outcomes | Run-in end (Day 0), Intervention end (Day 28), Follow-up end (Day 35)
  Psychological and behavioral outcomes will be assessed using multiple validated questionnaires. Each scale will be reported and analyzed separately: Diabetes Distress Scale (DDS): 17 items, scored 1-6; higher scores indicate greater distress; General Self-Efficacy Scale (GSES): 10 items, scored 1-4, total 10-40; higher scores indicate stronger self-efficacy; WHO-5 Well-Being Index: 5 items, raw score 0-25 transformed to 0-100; higher scores indicate better well-being; Summary of Diabetes Self-Care Activities (SDSCA): Items scored 0-7 days per week; higher scores indicate better diabetes self-management behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China